CLINICAL TRIAL: NCT01576822
Title: Complementary and Alternative Medicine Detoxification: Safety and Efficacy
Brief Title: Sauna Detoxification Study: Pilot Feasibility
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bastyr University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: H35B11; 4R00AT004711-03 (NIH)
Record Dates: First submitted 2012-02-01; First posted 2012-04-13 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-10

CONDITIONS: Hyperthermia
Keywords: Detoxification; Sauna
MeSH Terms: conditions — Hyperthermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low Dose (Active Comparator): Participants randomized to this group will undergo a protocol consisting of 1 hour of sauna therapy per day, for a minimum of 3 days per week, completed in 3 weeks or less (21 days). (9 total sessions, 9 hours of sauna). Participants will be able to schedule visits on any of 7 days per week. Maximum flexibility in hours of operation as well as flexibility in which days are attended will be utilized to increase likelihood of retention. Participants will be able to attend 9 consecutive sessions, should they wish.
  Interventions: Other: This protocol will utilize a sauna as the primary method of detoxification.
- High Dose (Active Comparator): Participants randomized to this group will undergo a protocol consisting of 2 hours of sauna therapy per day, for a minimum of 5 days per week, completed in 3 weeks or less (21 days). (15 total sessions, 30 hours of sauna). Participants will be able to schedule visits on any of 7 days per week. Maximum flexibility in hours of operation as well as flexibility in which days are attended will be utilized to increase likelihood of retention. A participant may attend visits for 15 consecutive days, should they wish.
  Interventions: Other: This protocol will utilize a sauna as the primary method of detoxification.

INTERVENTIONS:
Other: This protocol will utilize a sauna as the primary method of detoxification. — This study is a randomized, 2-arm, dose-finding safety and feasibility trial. After screening, informed consent and randomization, participants will complete a medically-monitored sauna-based detoxification program.
  High Dose Participants randomized to this group will undergo a protocol consisting of 2 hours of sauna therapy per day, for a minimum of 5 days per week, completed in 3 weeks or less (21 days). (15 total sessions, 30 hours of sauna).
  Low Dose Participants randomized to this group will undergo a protocol consisting of 1 hour of sauna therapy per day, for a minimum of 3 days per week, completed in 3 weeks or less (21 days). (9 total sessions, 9 hours of sauna).

SUMMARY:
The goal of this study is to assess the feasibility of the approach, conduct a dose-finding investigation, and obtain pilot data on hyperthermia via sauna to apply in follow-up trials in the assessment of human chemical body burden reduction, for general wellness, detoxification, and pain reduction.

The investigators wish to determine if a hyperthermia-based detoxification protocol is feasible to conduct: including assessment of recruitment, enrollment, retention, protocol adherence, adverse events, and changes in serum polychlorinated biphenyls (PCBs).

DETAILED DESCRIPTION:
According to our nationwide survey of Naturopathic Physicians regarding use of detoxification, approximately 80 percent of NDs (Naturopathic Doctors) use some type of detoxification interventions in clinical practice on a regular basis. Of the interventions used, 66% of respondents reported using sauna therapy. Of the conditions treated, over 80 percent of practitioners use sauna-based detoxification for "general cleansing/preventive medicine." This protocol will utilize a sauna as the primary method of detoxification.

Previous studies on hyperthermia-based protocols for detoxification have been methodologically challenged and are not readily reproducible. Furthermore, there are no studies in the literature that identify how long of a protocol is tolerated, is feasible in the general population, or how long is needed to observe PCB (or other pollutant reduction). Therefore, we will employ a "high-dose" protocol and a "low-dose" protocol, based on ranges reported in the literature, in order to evaluate dose-finding outcomes to hyperthermia, including tolerability, retention, and participant-reported outcomes.

High Dose Participants randomized to this group will undergo a protocol consisting of 2 hours of sauna therapy per day, for a minimum of 5 days per week, completed in 3 weeks or less (21 days). (15 total sessions, 30 hours of sauna). Participants will be able to schedule visits on any of 7 days per week. Maximum flexibility in hours of operation as well as flexibility in which days are attended will be utilized to increase likelihood of retention. A participant may attend visits for 15 consecutive days, should they wish.

Low Dose Participants randomized to this group will undergo a protocol consisting of 1 hour of sauna therapy per day, for a minimum of 3 days per week, completed in 3 weeks or less (21 days). (9 total sessions, 9 hours of sauna). Participants will be able to schedule visits on any of 7 days per week. Maximum flexibility in hours of operation as well as flexibility in which days are attended will be utilized to increase likelihood of retention. Participants will be able to attend 9 consecutive sessions, should they wish.

ELIGIBILITY:
Inclusion Criteria:

1. 21-35 years.
2. Body mass index (BMI) 19 to 30 kg/m2 at the screening evaluation.
3. Ability to schedule and attend daily visits for the duration of the study.
4. If female, willingness to use barrier contraception (e.g., cervical cap, diaphragm, condom, metal IUD (non- hormone)) throughout the study and take a pregnancy test at screening, and weekly during the study.

Exclusion Criteria:

1. Pregnant, or trying to become pregnant in the three months following screening.
2. Current use of any prescribed pharmaceutical medications (including oral contraceptive pills, without additional barrier contraception).
3. Participants who have a BMI greater than 30 kg/m2, elevated fasting blood sugar, bradycardia, hyper or hypotension or evidence of a medical condition.
4. A diagnosis of any chronic medical condition (e.g., multiple sclerosis, diabetes, or endocrine disorders, liver disease, kidney disease, HIV/AIDS, or cancer, or with a reported history of substance abuse or mental illness within the past 5 years, or a mental health disorder in the past 6 months.
5. Clinical chemistry lab values outside of reference lab normal ranges (except in cases of ranges within 10% ULN and isolated measurements in the absence of chronic disease).
6. Recent infection (<14 days), open sores, or communicable skin conditions.
7. Current use of any tobacco products or illicit drugs.
8. Any condition that in the opinion of the investigators or IRB would preclude the safe completion of the study (e.g., clinical or mental health concerns that arise from the screening questionnaire or physical exam).

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2011-11; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Recruitment/Retention | Up to 6 months
  Assess recruitment/retention goals/milestones
Protocol adherence | Up to 6 months
  Assess protocol adherence
Change from baseline in Clinical Chemistry Panel | Baseline and 4 weeks
  Complete metabolic panel, within normal limit (y/n)?
AE Monitoring | Up to 6 months
  Adverse event monitoring tool: FDA Monitoring of Side Effects System (MOSES)
Vital signs | Up to 6 months
  Vital signs within normal limits (y/n)?
Participant-reported outcome questionnaire | Baseline and up to 4 weeks
  NIH PROMIS Questionnaire
Short Form 36 health survey | Basleine and up to 4 weeks
  Health survey questionnaire

SECONDARY OUTCOMES:
Polychlorinated biphenyls | Baseline and 4 weeks
  Measure serum concentrations of PCBs

CONTACTS AND LOCATIONS:
Overall Officials: Jason Allen, N.D., MPH, Principal Investigator — Bastyr University
Locations (1):
- Bastyr University Clinical Research Center, Kenmore, Washington, United States